CLINICAL TRIAL: NCT02559219
Title: Smart Adult Living After Childhood Cancer (SmartALACC) Online Care Plans: Feasibility and Patient Satisfaction
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 36914
Record Dates: First submitted 2015-06-23; First posted 2015-09-24 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Childhood Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Questionniares

SUMMARY:
Smart Adult Living After Childhood Cancer (SmartALACC) Online Care Plans: Feasibility and Patient Satisfaction is a pilot project designed to test the feasibility and acceptability of use of an online care plan generator for adult survivors of pediatric cancers.

Because of improvements in cancer screening, diagnosis and treatment, there are an estimated 13 million cancer survivors living in the U.S. today, with projected growth to 18 million by 2020 (De Moor). These survivors include survivors of leukemia and lymphoma, as well as solid tumors including breast, colon, testicular and prostate cancers. It also include a subset of patients who are survivors of pediatric cancers, as over 80% of children diagnosed with cancer today are cured. In fact, it is estimated that 1 in every 600 young adults between the ages of 20-35 is a cancer survivor (Dreyer, Hewitt, Greenlee).

Cancer patients as a whole, despite improved cure rates, have been shown to receive inadequate medical care as survivors. Comprehensive survivorship care should include routine age appropriate medical care as well as information about prior diagnosis and treatment, and screening for recurrence of their primary malignancy as well as secondary malignancies, and screening for late effects of cancer treatment (Earle, Craig). Adult survivors of pediatric cancer, exposed to life-saving but toxic treatments during times of growth and development, are particularly prone to late effects but also have been shown to have inadequate monitoring and follow up. This is a concern as late effects of treatment are sometimes silent for years or decades after completion of cancer therapy and that adult survivors of childhood cancer, years from their diagnosis and treatment, have been shown to have alarming rates of life threatening chronic health conditions compared to their peers (Oeffinger). Thus, these late effects may emerge during adulthood when patients have moved on from the care of their primary oncologist. Complicating matters, primary care providers, who often assume the care of these patients, may not have the knowledge or tools necessary to appropriately care for survivors of childhood cancer (Suh).

National organizations have come together to identify ways to improve quality of and access to long term follow up care for adult survivors of childhood cancer. The Children's Oncology Group published Long Term Follow up guidelines which recommend lifelong risk based follow up care and screening (COG guidelines). In addition, in 2005, the Institute of Medicine published a report, From Cancer Patient to Cancer Survivor: Lost in Transition gave recommendations to improve health outcomes of cancer survivors which includes the receipt of a comprehensive care summary and follow up plan to aid in appropriate risk based follow up care (Hewitt). Despite these recommendations childhood cancer survivors knowledge about past diagnosis and treatment and engagement in follow up care is suboptimal (Kaden-Lottick, Nathan). It has been demonstrated that pediatric cancer survivors are not receiving care summaries, and thus may try to find appropriate follow up information via the other sources such as the internet (Casillas).

Oncolife, a free online tool to create survivorship care plans, was created in May 2007 (Hill 2009), and has been housed at maintained at the University of Pennsylvania since then. This tool has shown to be feasible way to provide information and care plans to survivors of adult cancers. In addition, survivors who have used the resource, state that it will, or has already, positively influenced communication about cancer related follow up with their healthcare team (Hill 2013).

The study aim is to adapt Oncolife to provide individualized information for adult survivors of childhood cancer with the unique recommendations for long term follow up for pediatric cancer survivors. Oncolife has already been collecting data on plans created by adult survivors of adult cancers and has been reviewed by the IRB previously (IRB#806368 and #811528 note: previously called Oncolink). Adaption of Oncolife to meet the needs of adult survivors of childhood cancer will improve access to high quality electronic health information as patients may find long term follow up guidelines cumbersome or largely irrelevant to their needs depending on their specific exposures. Individualizing the available information to a particular survivor will allow for better understanding of and improved adherence to recommended cancer related follow up care. We propose to develop survivorship care plans in a way that will most benefit users, thus after creation of the Smart Adult Living After Childhood Cancer care plan we will ask for patient input via survey immediately after receipt of their care plan and in a one month follow up survey.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a cancer diagnosis of acute lymphoblastic leukemia or Hodgkin's lymphoma
2. Diagnosis before age 21 years
3. Currently off therapy and considered in remission
4. Currently 15 years or older

Exclusion Criteria:

1. Persons who have never had cancer or who have another pediatric malignancy (Wilms tumor, neuroblastoma) as the website will not yet be adapted to create care plans for them.
2. Persons who were diagnosed with cancer >21 years. This program is designed for survivors of pediatric cancers. Survivors of adult cancers are referred to the existing information provided by Oncolink, Oncolife and the LIVESTRONG survivorship care plans.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: any person who has received a cancer diagnosis of acute lymphoblastic leukemia (ALL) or Hodgkins lymphoma (HL) before the age of 21 and now is 15 years or older and is now off therapy (considered in remission).
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-12; Primary Completion 2016-09 (Actual); Study Completion 2016-09-16 (Actual)

PRIMARY OUTCOMES:
Number of subjects completing questionnaires | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Christine Hill-Kayser, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States